CLINICAL TRIAL: NCT00176904
Title: Treatment of Lysosomal and Peroxisomal Inborn Errors of Metabolism by Bone Marrow Transplantation
Brief Title: Stem Cell Transplant for Inborn Errors of Metabolism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT1995-01; NCT00005894 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Adrenoleukodystrophy; Metachromatic Leukodystrophy; Globoid Cell Leukodystrophy; Gaucher's Disease; Fucosidosis; Wolman Disease; Niemann-Pick Disease; Batten Disease; GM1 Gangliosidosis; Tay Sachs Disease; Sandhoff Disease
Keywords: Inborn errors; Storage disease; errors of metabolism; stem cell transplant
MeSH Terms: conditions — Adrenoleukodystrophy; Leukodystrophy, Metachromatic; Leukodystrophy, Globoid Cell; Gaucher Disease; Fucosidosis; Wolman Disease; Niemann-Pick Diseases; Neuronal Ceroid-Lipofuscinoses; Gangliosidosis, GM1; Tay-Sachs Disease; Sandhoff Disease | interventions — Stem Cell Transplantation; Bone Marrow Transplantation; Busulfan; Cyclophosphamide; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treated Patients (Experimental): All patients treated with protocol regimen (chemotherapy and surgery).
  Interventions: Procedure: Stem Cell Transplant; Drug: Busulfan, Cyclophosphamide, Antithymocyte Globulin

INTERVENTIONS:
Procedure: Stem Cell Transplant — The purpose of hematopoietic cell transplantation is to introduce hematopoietic cells from a normal donor that contains an enzyme able to get rid of the substances that have accumulated in the body of patients with storage diseases. Hematopoietic cells can come from bone marrow, peripheral blood (i.e., the blood circulating in our body's blood vessels) or umbilical cord blood (i.e., blood taken from the umbilical cord after a baby is born and umbilical cord is cut).
  Other Names: Bone marrow transplant
Drug: Busulfan, Cyclophosphamide, Antithymocyte Globulin — Subjects will receive BUSULFAN intravenously (IV)- patients < or= 12 kg 1.1 mg/kd/dose IV every 6 hours for 16 doses; patients > 12kg 0.8 mg/kg/dose IV every 6 hours for 16 doses - via the Hickman line four times daily for 4 days, CYCLOPHOSPHAMIDE intravenously (50 mg/kg/day IV over 2 hours) via the Hickman line once a day for 4 days, and ANTI-THYMOCYTE GLOBULIN IV (15 mg/kg/day over 2 hours) via the Hickman line twice daily for three days before the transplant. These three drugs are being given to help the new marrow "take" and grow. METHYLPREDNISOLONE will be given as a pre-medication for the ATG.
  Other Names: Busulfex, Cytoxan, ATG

SUMMARY:
The purpose of this study is to determine the safety and engraftment of donor hematopoietic cells using this conditioning regimen in patients undergoing a hematopoietic (blood forming) cell transplant for an inherited metabolic storage disease.

DETAILED DESCRIPTION:
Prior to transplantation, subjects will receive Busulfan intravenously (IV) via the Hickman line four times daily for 4 days, Cyclophosphamide intravenously via the Hickman line once a day for 4 days, and Anti-Thymocyte Globulin (ATG) intravenously (IV) via the Hickman line twice daily for three days before the transplant. These three drugs are being given to subjects to help the new marrow "take" and grow.

On the day of transplantation, the donor's hematopoietic cells will be transfused via central venous catheter.

After hematopoietic cell transplant, subjects will then receive two drugs, cyclosporin and either methylprednisolone or Mycophenolate Mofetil (MMF). Cyclosporin and methylprednisolone or MMF are given to help prevent the complication of graft-versus-host disease and to decrease the chance that the new donor cells will be rejected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adrenoleukodystrophy, metachromatic leukodystrophy, globoid cell leukodystrophy, Gaucher's disease, Fucosidosis, Wolman disease, Niemann-Pick disease and Batten disease (CLN3) who have a human leukocyte antigen (HLA)-identical or haplotype mismatched (at 1-3 antigens) related marrow, or umbilical cord blood donor. One or two umbilical cord blood (UCB) units may be used.
* Patients with GM1 gangliosidosis, Tay Sachs disease or Sandhoff disease who have a HLA-identical or 1 antigen mismatched related or unrelated donor, or suitably matched umbilical cord blood unit(s). One or two UCB units may be used.
* Patients with adrenoleukodystrophy must have magnetic resonance imaging (MRI) findings, neurological and neuropsychometric function consistent with the diagnosis, and for boys with parietal-occipital dysmyelination a performance intelligence quotient (IQ) ≥80. In cases, when the performance IQ is not ≥80, the protocol committee may recommend transplant if the patient's clinical condition and neuropsychometric status are deemed to be acceptable based upon consideration of such factors as age at onset of cerebral disease, magnitude of change in performance IQ and neurologic deficits.
* Patients with arylsulfatase A deficiency (Metachromatic Leukodystrophy) must have either the presymptomatic late infantile, juvenile or adult form of the disease and must have acceptable neurological and neuropsychometric function.
* Patients with galactocerebrosidase deficiency (Globoid Cell Leukodystrophy) must have acceptable neurological and neuropsychometric function.
* Patients with acid lipase deficiency (Wolman disease) must have a liver biopsy that documents no evidence of hepatic cirrhosis, and acceptable neurological and neuropsychometric function.
* Patients with fucosidase deficiency (Fucosidosis) must have acceptable neurological and neuropsychometric function.
* Patients with glucocerebrosidase deficiency (Gaucher's Disease) must have acceptable neurologic and neuropsychometric function.
* Patients with Batten's disease (CLN3) must have acceptable Neurological and neuropsychometric function.
* Absence of major organ dysfunction. Organ evaluation results as follows:
* Cardiac: ejection fraction >30%
* Renal: serum creatinine <2x normal or creatinine clearance 60 mL/min.
* Hepatic: total bilirubin <2x normal and Aspartate aminotransferase (AST) <2x normal
* Signed consent.

Exclusion Criteria:

* Patients with symptomatic late infantile form of metachromatic leukodystrophy.
* Patients with symptomatic infantile globoid leukodystrophy.
* Note: Patients with Hurler syndrome, mucopolysaccharidosis (MPS) VI, or Mannosidosis disease are no longer eligible for this protocol, but can be transplanted under protocol MT 9907 (NCT00176917 - Hematopoietic Cell Transplantation for Hurler Syndrome, Maroteaux Lamy Syndrome (MPS VI), and Alpha Mannosidase Deficiency (Mannosidosis)).
* Pregnancy
* Evidence of human immunodeficiency virus (HIV) infection or known HIV positive serology
* Patients or parents are psychologically incapable of undergoing bone marrow transplant (BMT) with associated strict isolation or documented history of medical non-compliance.
* Patients ≥ 50 kg may be at risk for having cell doses below the goal of ≥ 10 x 10^6 CD34 cells/kg and therefore will not be eligible to receive unrelated peripheral blood stem cells (PBSCs)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 1995-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Orchard, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Miller WP, Rothman SM, Nascene D, Kivisto T, DeFor TE, Ziegler RS, Eisengart J, Leiser K, Raymond G, Lund TC, Tolar J, Orchard PJ. Outcomes after allogeneic hematopoietic cell transplantation for childhood cerebral adrenoleukodystrophy: the largest single-institution cohort report. Blood. 2011 Aug 18;118(7):1971-8. doi: 10.1182/blood-2011-01-329235. Epub 2011 May 17. PMID 21586746

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Treated With Stem Cell Transplant: All patients treated with protocol regimen (chemotherapy and stem cell transplant).
Period: Overall Study
Arm/Group | Patients Treated With Stem Cell Transplant
Started | 135
Completed | 135
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Treated With Stem Cell Transplant
Number analyzed (Participants) | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 117
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 91
Region of Enrollment [Number; unit: participants]
  United States | 135

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of patients alive at designated timepoints after transplant.
Time Frame: 100 Days, 1 Year and 3 Years
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Stem Cell Transplant
Number analyzed (Participants) | 135
Participants
  Day 100 | 120
  1 Year | 92
  3 Years | 81

2. Secondary Outcome: Overall Donor Engraftment
Description: Number of patients with full donor chimerism (state in bone marrow transplantation in which bone marrow and host cells exist compatibly without signs of graft-versus-host rejection disease) by Day 100 post-transplant of at least 90%.
Time Frame: Day 100
Population: 1 Patient not included due to early death (before day 40).
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Stem Cell Transplant
Number analyzed (Participants) | 134
Participants | 123

3. Secondary Outcome: Number of Patients With Grade II-IV Acute Graft-Versus-Host Disease
Description: Number of patients who exhibited acute graft-versus-host disease by Day 100 post transplant. Graft-versus-host disease (GVHD) is a complication that can occur after a stem cell or bone marrow transplant in which the newly transplanted material attacks the transplant recipient's body. Grade I=mild, Grade II=moderate, Grade III=severe, Grade IV=life threatening.
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Stem Cell Transplant
Number analyzed (Participants) | 135
Participants | 34

4. Secondary Outcome: Number of Patients With Grade III-IV Acute Graft-Versus-Host Disease
Description: as for outcome 3
Time Frame: Day 100
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Stem Cell Transplant
Number analyzed (Participants) | 135
Participants | 13

5. Secondary Outcome: Number of Patients With Chronic Graft-Versus-Host Disease
Description: Number of patients who exhibited chronic graft-versus-host disease by 1 Year post transplant. Graft-versus-host disease (GVHD) is a complication that can occur after a stem cell or bone marrow transplant in which the newly transplanted material attacks the transplant recipient's body. Chronic GVHD is an extension of this syndrome.
Time Frame: 1 Year Post Transplant
Measure: Number; unit: Participants
Arm/Group | Patients Treated With Stem Cell Transplant
Number analyzed (Participants) | 135
Participants | 13

ADVERSE EVENTS:
Time Frame: Serious adverse experiences were collected during the first 100 days after transplant then 6 months and annually for 3 years.
Description: Selected serious adverse experiences (graft failure/autologous recovery, severe acute GVHD (grades III and IV) and death were collected during the first 100 days after transplant then 6 months and annually for 3 years. After day 100, only death or an unexpected adverse event will be reported. Adverse events were not collected in this study.
Arm/Group | Patients Treated With Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 62/135
Other Adverse Events (participants affected / at risk) | 0/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Treated With Stem Cell Transplant (N=135)
Auto recovery (General disorders) | 9 (9) — Delayed side effects that includes, loss of appetite, nausea and vomiting, changes in vision, mouth and throat soreness, diarrhea, difficulty sleeping and fatigue, infection, hair loss, skin reactions and graft-versus-host disease.
Death (General disorders) | 54 (54)
Primary graft failure (Blood and lymphatic system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Change in Neuropsychometric function data is not available. Data would have been noted as descriptive and patient specific, as well as disease specific; not table format. No formal analysis was intended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No